CLINICAL TRIAL: NCT02155517
Title: Phase 4: CLINICAL EVALUATION OF TWO PHARMACOKINETICS MODELS OF PROPOFOL IN HEALTHY PEOPLE
Brief Title: Clinical Effect of Two Pharmacokinetics Model of Propofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tiva Group (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Carolina Frederico, Anestesiologo, Tiva Group
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 019CBCEA032013
Record Dates: First submitted 2014-05-19; First posted 2014-06-04 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: TCI,Schnider Model, Cortinez Model, BIS, Cardiac Output.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol Infusion (Experimental): Propofol will be administered using a commercially available target-controlled infusion with an incorporated pharmacokinetic model developed by Schnider and Cortinez (arcomed ag, Medical System, Switzerland )..
  The study will make in two stages:
  STAGE I: All volunteers will receive propofol infusion with the first model randomly chosen (Schnider or Cortinez) using TCI device, and the initial effect-site target concentration of propofol will be 3 ug/ml for 20 minutes.
  STAGE II: 72 hours after stage I . All volunteers will receive propofol infusion with the first model randomly chosen (Schnider or Cortinez) using TCI devices, and the initial effect-site target concentration of propofol will be 3 ug/ml for 20 minutes.
  Interventions: Drug: Evaluation of propofol effect

INTERVENTIONS:
Drug: Evaluation of propofol effect — The study will make in two stages:
  STAGE I: All volunteers will receive propofol infusion with the first model randomly chosen (Schnider or Cortinez) using TCI device, and the initial effect-site target concentration of propofol will be 3 ug/ml for 20 minutes.
  Other Names: Propofol Induced sedation
Drug: Evaluation of propofol effect — STAGE II: 72 hours after stage I . All volunteers will receive propofol infusion with the first model randomly chosen (Schnider or Cortinez) using TCI devices, and the initial effect-site target concentration of propofol will be 3 ug/ml for 20 minutes.
  Other Names: Propofol Induce sedation

SUMMARY:
Actually, Schnider and Cortinez models represent pharmacokinetics models of propofol more complete published until now. Schnider was derived from 24 healhty people, and including other covariates in addition to weight, such as age, height and lean body mass though. Schnider model should not be used in obese patients. Cortínez model was derived from 20 obese patients. The differences between both models has been founded at the initial drug distribution, that means V1 and the constant Ke0 ( pharmacokinetics factors that define the plasma-effect equilibration time). We believe that Cortinez model also could be used in No OBESE patients because is an allometric model, and one way to evaluate and to compare both pharmacokinetics models is studying the temporary course of the effect.

The main objective of our study is to evaluate BIS and Cardiac Output values during propofol-induced sedation using Schnider and Cortinez models in Target Controlled infusion in non obese healthy volunteer.

DETAILED DESCRIPTION:
The study was approved by the ethics committee of the Avila Clinic. After informed consent, 10 volunteers aged 18-60 años, ASA I, Body mass Index < 30 were included.

The patients fasted for 8h before the protocol and they will not receive premedication. After arrival in the operating room, and insertion of 18-gauge intravenous cannulas placed into the forearm, a Ringer's lactate solution will be initiated. Oxygen therapy at a rate of 5 litres per minute will be administered in spontaneous ventilation. In case of hypoventilation (saturation (SaO2) <95% manual ventilation with a mask at 10 l/min of O2 will be administered. All volunteer will be monitoring with EKG, Blood pressure, Pulse Oximetry, Bispectral Index and Cardiac output.

Propofol will be administered using a commercially available target-controlled infusion with an incorporated pharmacokinetic model developed by Schnider and Cortinez (arcomed ag, Medical System, Switzerland ). Each volunteer will be studied twice, that means which each subject then acts as their own control.

The study will make in two stages:

STAGE I: All volunteers will receive propofol infusion with the first model randomly chosen (Schnider or Cortinez) using Target Controlled Infusion device, and the initial effect-site target concentration of propofol will be 3 ug/ml for 20 minutes.

STAGE II: 72 hours after stage I . All volunteers will receive propofol infusion with the first model randomly chosen (Schnider or Cortinez) using Target Controlled Infusion devices, and the initial effect-site target concentration of propofol will be 3 ug/ml for 20 minutes.

Lost of consciousness will be evaluated by an independent observer using two different criteria: OAA/S score <2 (OAA/S2) corresponding to the absence of response to moderate prodding and loss of eyelash reflex (LOER). Time to OAA/S2 and time to LOER will be measured as well as corresponding brain and plasma concentrations of propofol. At the same time, BIS and Cardiac output values will be recording.

After 20 minutes, the infusion will be stopped. Recovery of consciousness (ROC), which will be assessed every 10s until patients wake up, and the values of Ce, BIS and Cardiac Output.

The electroencephalogram (EEG) activity will be monitored by BIS Quatro platform® electrodes and a BIS VISTA™ 1.01 monitor Vista the bispectral index (Covidien, USA). The information will be recording every 20 seconds The cardiac output will be measured using Monitor ICON ® Electrical Cardiometric ™

Arterial blood pressure, heart rate, SaO2, respiratory frequency will be measured before to start propofol infusion and then every 3 minutes until the end of trial. A decrease in systolic arterial pressure ≥30 % of the basal value will be considered as hypotension, and heart rate <45 defined bradycardia.

STATISTICAL ANALYSIS This is a prospective, descriptive and comparative study. We will use the Wilcoxon-Mann-Whitney nonparametric test applied for two independent samples

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I
* Aged 18-60 years
* Patients with Body mass Index < 30.

Exclusion Criteria:

* Patients with Body mass Index > 30.
* Patients presenting psychiatric or neurological disorders , endocrine-metabolical problems, respiratory and cardiac diseases, or with allergies problems.
* Patients who are pregnant or breastfeeding.
* Patients treated with psychotropic drugs, including alcohol, in the 48 hours prior.
* Patients with previous history of anesthetics complications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sedation Levels | During propofol infusion period
  We will use Ramsey Sedation Scale to evaluate LOC at the beginning of the infusion and after 20 minutes we will evaluate the recovery of consciousness after the infusion is stopped.

SECONDARY OUTCOMES:
Bispectral index values | During a propofol infusion period
  We will use BIS monitor (BIS Vista, Covidien). The data will be collected in excel data sheet
Hemodynamics values | During propofol infusion period
  We will measure cardiac output using Monitor ICON ® Electrical Cardiometric ™, every 3 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Ramirez, Dr, Principal Investigator
Locations (1):
- Clinica Avila, Caracas, Distrito Federal, Venezuela